CLINICAL TRIAL: NCT04935372
Title: β-AARC: Cohort Study for the Identification of Blood-based Biomarkers in a Population With Subjective Cognitive Decline
Acronym: β-AARC
Status: Active, not recruiting | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: β-AARC_BBRC2021
Record Dates: First submitted 2021-06-08; First posted 2021-06-23 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Preclinical Alzheimer; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjective cognitive decline: Male and female, aged 55 to 80 years with subjective cognitive decline, either cognitively unimpaired or with mild cognitive impairment
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Cross sectional analyses The two main variables for the analysis will be: Values of biomarker concentrations in blood and their correlations with CSF biomarkers and the development of prodromal AD for the cognitively unimpaired SCD population. Other variables of interest for the study are, among others, risk factors, cognitive status, measurements of brain structure and function, mental health, chronic diseases, environmental exposures, age and sex.
  Longitudinal analyses Longitudinal analyses will estimate the association between the intensity of the subjective complaint and the rate of progression between the diagnostic categories; The association of biomarkers, risk factors and other clinical variables with the rate of progression between the diagnostic categories; The association of cognitive and neuroimaging variables with the rate of progression between the diagnostic categories; The evolution of the complaint itself and its relation to the other variables described.

SUMMARY:
The overall (cross-sectional) objective of this study is to detect and describe the profile of AD-related blood biomarkers in a population with SCD (including individuals with MCI) with the ultimate goal of investigating their capacity to predict underlying AD pathology. Longitudinally, the β-AARC_BBRC2021 study fundamentally aims at assessing the ability of AD-related blood-based biomarkers to predict disease progression in the Alzheimer's continuum.

To achieve these cross-sectional and longitudinal objectives, an exhaustive set of clinical, risk factors, cognitive, mental health and neuroimaging data will be collected, as well as blood and CSF samples, from which AD-related fluid biomarkers will be determined.

As a secondary objective, we will investigate the efficacy and accuracy of the Altoida NMI as a novel digital biomarker for identifying patients with SCD or MCI that have underlying AD pathology (cross-sectionally) and to test the capacity of the Altoida NMI to track disease progression in these popoulations (longitudinally).

ELIGIBILITY:
Inclusion Criteria:

1. Cognitively unimpaired persons with SCD as well as individuals with MCI.
2. To sign the study informed consent form, approved by the corresponding authorities.
3. Participation (in-person at the institution or telephonically) of a relative to inform on the participant subjective memory decline and on the clinical interview*.
4. Men and women between 55 and 80 years old
5. Memory Alteration Test (M@T) ≤45
6. Good knowledge of the either Spanish or Catalan language and being literate.

Exclusion Criteria:

1. Presence of clinically relevant psychiatric disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) criteria: major depressive disorder, generalized anxiety disorder, schizophrenia and bipolar disorder, or any other condition that might impact cognition or performance on cognitive assessments as judged by the investigator
2. Parkinson's disease, epilepsy in treatment and with frequent seizures (> 1 / month) in the last year, multiple sclerosis or other neurodegenerative disease.
3. Contraindication to perform an MR scan: claustrophobia, pacemaker, metallic implants, etc.
4. Contraindication to lumbar puncture
5. Acquired brain injury: history of cranioencephalic trauma with gross parenchymal or extra axial lesion, hemorrhagic ischemic stroke, brain tumors and other aetiologies that can cause acquired brain damage (chemotherapy or brain radiotherapy).
6. Investigator's criteria: Subjects that show any condition that, in the opinion of the investigator, could interfere in the proper execution of the study procedures and / or in their future permanence in the study.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two-hundred participants, aged 55 to 80 years with subjective cognitive decline, will be primarily selected from the population seeking medical advice on their cognitive performance to Primary care units. In addition, other conventional recruitment strategies may be used (e.g. participants of ongoing or ended BBRC-sponsored studies,novel recruitment calls…).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
CSF Aβ42/Aβ40 ratio | Through study completion, an average of 1 year
  The capacity of plasma biomarkers to predict (alone or in combination of covariates) Alzheimer's pathology

SECONDARY OUTCOMES:
Cost effectiveness | Through study completion, an average of 1 year
  The ratio between the cost and predictive capacity of these variables will be considered to derive a triaging algorithm for primary care

CONTACTS AND LOCATIONS:
Locations (1):
- BarcelonaBeta Brain Research Center, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided